CLINICAL TRIAL: NCT03318510
Title: Laser Speckle Flowgraphy in Patients With Normal Tension Glaucoma - a Pilot Study
Brief Title: LSFG in Patients With Normal Tension Glaucoma Tension Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Augenabteilung Allgemeines Krankenhaus Linz (Other)
Responsible Party: Principal Investigator, Matthias Bolz, Prof., Augenabteilung Allgemeines Krankenhaus Linz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AO Form 01-05/1.0
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Laser Speckle Flowgraphy — A commercially available LSFG system (LSFG-NAVI; Softcare Co., Ltd., Fukuoka, Japan) will be used in the present study. The LSFG device consists of a fundus camera equipped with a diode laser with a wavelength if 830 nm and charge-coupled device.

SUMMARY:
Glaucoma is the second leading cause of blindness worldwide. Literature shows increasing evidence that dysfunction of ocular microcirculation in the optic nerve influences the progression of glaucoma. Laser speckle flowgraphy (LSFG) represents a non-invasive method to quantify ocular perfusion also at the ONH. LSFG enables noninvasive quantification of microcirculation of the optic disc in Japanese glaucoma patients

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women aged over 50 years
* Subject is generally healthy with no current significant or a history of a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, metabolic, rheumatic, autoimmune, hematological or renal disorder, as determined by the investigator's clinical judgment through collection of medical history and performance of a physical examination. A significant disorder is defined as a disease or medical condition associated with impaired health status, requiring regular or current medical treatment and/or follow up. For the purposes of this study, an investigator may classify a medical condition as a nonsignificant disorder despite the fact that the subject receives treatment. Subjects having controlled Stage 1 hypertension (blood pressure of 140-159 mmHg systolic and/or 90-99 mmHg diastolic) are eligible for participation in this study
* Normal open angle in a gonioscopic examination
* Presence of glaucomatous optic disc changes in biomicroscopy and
* Visual field defects in at least two visual field examinations (Reliability criteria: fixation errors < 20%, false positives < 15%, and false negatives < 33%) Or
* Abnormal circumpapillary retinal nerve fiber layer thinning (RNFL evaluated by OCT)

Exclusion Criteria:

* History of ocular or systemic disease causing optic nerve damage
* History of IOP greater than 21 mm Hg (corrected by CCT)
* Participation in a clinical trial in the 3 weeks preceding the study
* Ocular surgery (including intravitreal injection) during the 3 months preceding the study
* Ametropia > 6 Dpt
* Smoking
* pre- or perimenopausal women
* Relevant ophthalmic diseases/conditions that could interfere with LSFG measurements (e.g. optic nerve head drusen, tilted disc, etc.)
* Opacities of the cornea (e.g. corneal scars, corneal oedema), the lens (e.g. LOCS-II grading > 2, posterior capsule opacification) or the vitreous (e.g. vitreous haemorrhage, asteroid hyalosis)
* Patients who are not able to cooperate or with insufficient ability to fixate (tremor, nystagmus)
* Blood donation in the 3 weeks preceding the study
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Ocular infection or clinically significant inflammation
* Pregnancy, planned pregnancy or lactating

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-20 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean blur ratio (LSFG) | 4 seconds

SECONDARY OUTCOMES:
Pulse-waveform parameters (LSFG) | 4 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- AKh Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No